CLINICAL TRIAL: NCT01449409
Title: Reduce IDentified UNcontrolled Asthma: A Real-time Randomized Administrative Outreach Study to Promote Asthma Guideline Implementation (RIDUNA)
Brief Title: Reduce IDentified UNcontrolled Asthma
Acronym: RIDUNA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert S. Zeiger, MD, PhD, Adjunct Physician Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB # 5808
Record Dates: First submitted 2011-10-03; First posted 2011-10-10 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Asthma
Keywords: Uncontrolled asthma; Asthma risk; Asthma impairment; Real time asthma outreach program
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Real-time asthma care outreach (Experimental)
  Interventions: Other: Real-time asthma care outreach

INTERVENTIONS:
Other: Real-time asthma care outreach — Real-time asthma care identification of uncontrolled asthma and real-time notification of patients and their physicians of uncontrolled asthma and directions to improve care. Patients without an asthma specialist visit in the prior 3 years are offered an expedited allergy department referral.
  Other Names: Expedited asthma care management
  Arms: Real-time asthma care outreach

SUMMARY:
The purpose of Reduce IDentified UNcontrolled Asthma (RIDUNA) is to determine the benefit of real-time identification of uncontrolled asthma by electronic administrative records linked to real-time notification of uncontrolled status to patients and asthma specialists with recommended guideline directed intervention by physicians. The investigators hypothesize that real-time outreach following National guideline asthma care recommendations, after real-time identification of an uncontrolled asthma event in persistent asthmatics on inhaled corticosteroids will lead to better improvements in asthma control (impairment and risk) compared to standard asthma care outreach.

DETAILED DESCRIPTION:
Co-primary Objectives: Determine the effectiveness of real-time identification administratively of uncontrolled asthma and real-time outreach administratively to optimize National asthma care guideline implementation compared to standard KP asthma outreach to improve asthma control (subsequent asthma impairment and risk, separately).

Hypothesis 1: Real-time notification of uncontrolled asthma status to asthma specialists and patients compared to standard Kaiser Permanente (KP) asthma outreach will reduce subsequent asthma impairment and risk, separately.

Hypothesis 2: Real-time notification of uncontrolled asthma status to asthma specialists and patients compared to standard KP asthma outreach will increase the proportion of patients who receive step-up care for impairment and risk.

Hypothesis 3: The real-time notification of uncontrolled asthma status to asthma specialists and patients compared to standard KP asthma outreach will lead to increased step-up care that will reduce subsequent asthma impairment and risk.

Hypothesis 4: Specific demographic characteristics (older age, female gender, non-Hispanic white ethnicity, higher census block education/income level) will be associated with a differential response in the intervention group.

Study Objectives:

1. Determine whether real-time notification of uncontrolled asthma status to asthma specialists and patients compared to standard KP asthma outreach will reduce subsequent asthma impairment and risk, separately.

2: Determine whether real-time notification of uncontrolled asthma status to asthma specialists and patients compared to standard KP asthma outreach will increase the proportion of patients who receive step-up care for impairment and risk.

3: Determine whether the real-time notification of uncontrolled asthma status to asthma specialists and patients will lead to increased step-up care that will reduce subsequent asthma impairment and risk compared to standard KP asthma outreach.

4: Determine whether there exist specific demographic characteristics (older age, female gender, non-Hispanic white ethnicity, higher census block education/income level) that are associated with a greater differential efficacy in the intervention group.

5. Determine in an exploratory analysis the frequency, characteristics (demographic, asthma severity, prior health care utilization, etc) and clinical outcomes (impairment and risk) of patients placed on omalizumab step-up therapy.

ELIGIBILITY:
Inclusion Criteria:

KPSC members at time of uncontrolled event:

1. 12-56 years of age
2. Continuously enrolled and with pharmacy benefit for the past year
3. Dispensed inhaled corticosteroid (ICS) in the past 6 months.
4. Uncontrolled asthma: defined within the past year

   * Impairment cohort: 7th short-acting beta-agonist (SABA) canister dispensed and/or
   * Risk (exacerbation) cohort: 2nd oral corticosteroid (OCS)dispensing with provider asthma exacerbation encounter within 2 days and at least 1 month after the first OCS dispensing.

Exclusion Criteria:

* Patients with chronic obstructive lung disease,
* emphysema,
* cystic fibrosis,
* chronic bronchitis,
* bronchiectasis,
* Churg Strauss,
* Wegener's,
* sarcoidosis,
* pulmonary hypertension or other clinically relevant non-asthma pulmonary disorder such as autoimmunity,
* immune deficiency,
* cancer,
* HIV,
* steroid dependent asthma,
* omalizumab therapy within the past 3 months, and
* requirement for an interpreter.

Ages: 12 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2011-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral corticosteroid courses for asthma exacerbations in risk cohort. | 1 year
  Measure in the follow-up year (1) frequency of patients requiring 2 or more oral corticosteroid courses in cohort with uncontrolled asthma based on risk
Short-acting beta-agonist dispensings. | 1 year
  Frequency of patients requiring 7 or more short-acting beta-agonist dispensings in cohort with uncontrolled asthma based on impairment.

SECONDARY OUTCOMES:
Frequency of patients with documented step-up care. | 1 year
Frequency, characteristics, and exacerbations of patients placed on omalizumab therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Zeiger, MD, PhD, Principal Investigator — Kaiser Permanente Southern California Region
Locations (1):
- Kaiser Permanente Southern California Region, San Diego, California, United States

REFERENCES:
- [Background] Zeiger RS, Schatz M, Li Q, Zhang F, Purdum AS, Chen W. Step-up care improves impairment in uncontrolled asthma: an administrative data study. Am J Manag Care. 2010;16(12):897-906. PMID 21348560
- [Background] Schatz M, Zeiger RS. Improving asthma outcomes in large populations. J Allergy Clin Immunol. 2011 Aug;128(2):273-7. doi: 10.1016/j.jaci.2011.03.027. Epub 2011 Apr 17. PMID 21497885
- See also: Kaiser Permanente Research and Evaluation Department Clinical Trials — http://www.kp-scalresearch.org/ClinicalTrials/ClinicalTrials.aspx
- See also: Kaiser Permanente Health Research — http://xnet.kp.org/newscenter/aboutkp/research-ctrs.html